CLINICAL TRIAL: NCT05731674
Title: Random Selection of Exercises Versus Self-Directed Training, for Laparoscopic Simulator Training - a Randomized Trial
Brief Title: Varied Practice on LAPSIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Responsible Party: Principal Investigator, Anishan Vamadevan, Research scholar, Bsc. in Medicine, Copenhagen Academy for Medical Education and Simulation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Varied Practice's on LAPSIM
Record Dates: First submitted 2022-06-30; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Skilss Acquisition for Virtual Reality Laparoscopic Training

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental)
  Interventions: Other: Random selection of excercises

INTERVENTIONS:
Other: Random selection of excercises — Participants in the intervention group will train using a random selection of excercises and complete the profiency-based traning program.
  Arms: Intervention

SUMMARY:
To investigate whether training using a random selection of exercises on a laparoscopic virtual reality simulator results in a stronger retention of skills when using a proficiency-based training program compared to conventional self-directed training.

ELIGIBILITY:
Inclusion Criteria:

* Medical Students enrolled at a Danish University

Exclusion Criteria:

* Not being enrolled at a medical program at a Danish University, having participated in other virtual reality studies regarding laparoscopy, have had training or practice in laparoscopy on either pigs or in the clinic, have any medical conditions that may hinder a standard learning process when it comes to skills acquisition (eg. parkinson's disease, limited eye-sight etc).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Time (minutes) to reach the predefined proficiency settings for the basic skills and the procedural module after 3-6 weeks without laparoscopic training. | 6 weeks

SECONDARY OUTCOMES:
Time (minutes) to reach the predefined proficiency settings for the basic skills | 6 weeks
  To examine any difference in training time for the two groups over-all
Time (minutes) to reach proficiency setting for the procedural module (salpingectomy due to an ectopic bleeding) | 6 weeks
  To examine if there is any difference in training time (minutes) for the two-groups when practicing on the procedural module (salpingectomy due to an ectopic bleeding)

CONTACTS AND LOCATIONS:
Locations (1):
- CAMES, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided